CLINICAL TRIAL: NCT01041963
Title: The Effect of Enalapril and Losartan on Peritoneal Membrane in Continuous Ambulatory Peritoneal Dialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Assist. Prf. Talerngsak Kanjanabuch, M.D / Department of nephrology, Division of Internal medicine, Faculty of medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 203/52
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Continuous Ambulatory Peritoneal Dialysis
Keywords: ACEI; ARB; CAPD; Peritoneal membrane transport
MeSH Terms: interventions — Enalapril; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Enalapril (Active Comparator)
  Interventions: Drug: Enalapril
- Enalapril plus Losartan (Active Comparator)
  Interventions: Drug: Enalapril plus Losartan
- Control (Placebo Comparator): Drug: antihypertensive agents, except ACE inhibitors and ARBs and spironolactone. Administration of antihypertensive agents will select as follows : CCB→β-blocker→α-blocker-->hydralazine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enalapril — Patients with hypertension will take 20-40mg enalapril per day, antihypertensive agents other than ACE inhibitors and ARBs and spironolactone will be allowed. Doses are adjusted appropriately to achieve and maintain the target blood pressure of 130/80 mmHg
  Other Names: Anapril
  Arms: Enalapril
Drug: Enalapril plus Losartan — Patients with hypertension will take 20-40mg enalapril plus 25-50mg losartan per day, antihypertensive agents other than ACE inhibitors and ARBs and spironolactone will be allowed. Doses are adjusted appropriately to achieve and maintain the target blood pressure of 130/80 mmHg
  Other Names: Anapril plus Loranta
  Arms: Enalapril plus Losartan
Drug: Placebo — Patients in the control group will administer antihypertensive agents, except ACE inhibitors and ARBs and spironolactone. Doses are adjusted appropriately to achieve and maintain the target blood pressure of 130/80 mmHg
  Other Names: Control
  Arms: Control

SUMMARY:
A prospective, randomized, open-label, Single-center clinical trial to determine whether Enalapril or Enalapril plus Losartan effect on Peritoneal membrane transportation.

DETAILED DESCRIPTION:
Detailed description:

Many peritoneal dialysis patients suffer from uremia due to inadequate dialysis or volume overload caused by failure of peritoneal membrane transport.One of the most important etiologies of peritoneal membrane failure are unavoidable to use high glucose-containing dialysate solution that induce injury to mesothelial cell.Previous data found that injured mesothelial cell produces Angiotensin (Ang) II to induce peritoneal inflammation and fibrosis. Blockade of the renin-angiotensin system by angiotensin-converting enzyme inhibition(ACEI) or angiotensin receptor antagonism (ARB) play a major role to slow this effect.

Although many trials in animal study have proved the benefit of ACEI and ARB in peritoneal membrane transport but clinical evidences in human are controversy. Up to now, all previous trials have limitation. First,The trials have small number of population(less than 20 in prospective randomized controlled trial). Second, The trials have multiple confounders on the study population because of the study include old case (that on peritoneal dialysis for many years) and new case (that just start treatment less than 1 year). Third, short duration of study(less than 3 months) to see the significant effect of RAAS blockade on peritoneal membrane transport. Forth, most study use dialysate albumin loss as an index of peritoneal membrane transport ,that less sensitivity to predict peritoneal membrane function. Fifth,no previous trials are attempted to study the effect of combination between ACEI and ARB. Therefore,we design to study the effect of both ACEI and ARB in a larger number of population, only in new case which are just recently found to be on peritoneal dialysis, our study is taken in longer duration and use both modified peritoneal equilibrium test and dialysate CA125 as an index of peritoneal membrane (physiology and anatomic index).This research will demonstrate efficacy of Enalapril and Losartan on Peritoneal membrane transportation lead to improve quality of life in CAPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. All patients received CAPD more than 1 months but less than 1 year
2. Subjects of either sex, more than 20 years old
3. Hypertension
4. Provision of written informed consent by subject or guardian

Exclusion Criteria:

1. No history of taking an ACE inhibitor or angiotensin-receptor blockers or aldosterone antagonist for at least 2 month
2. Serum potassium more than 5.5 mEq/L
3. History of renal artery stenosis
4. Peritonitis or volume overload within the preceding 1 month
5. Myocardial infarction within the preceding 6 months or clinically significant valvular disease or any active cardiovascular disease
6. History of malignant hypertension or hypertensive encephalopathy or cerebrovascular accident within the preceding 6 months
7. Any condition that may have precluded a patient from remaining in the study, such as alcohol or drug abuse, chronic liver disease, malignant disease, or psychiatric disorder
8. History of allergy or intolerance to an ACE inhibitor or ARB
9. Hypotension defined as systolic blood pressure less than 90 mmHg

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Change in dialysate CA-125 and modified peritoneal equilibrium test | 12 months

SECONDARY OUTCOMES:
Dialysis adequacy, residual renal function, hospitalization, peritonitis episodes, any adverse drug effects, death from any cause | every 1 month, except for dialysis adequacy evaluate every 3 mo

CONTACTS AND LOCATIONS:
Overall Officials: Talerngsak Kanjanabuch, Assist. Prf., Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn university, Bangkok, Thailand